CLINICAL TRIAL: NCT04394858
Title: A Prospective, Multi-Institutional Phase II Trial Evaluating Temozolomide vs. Temozolomide and Olaparib for Advanced Pheochromocytoma and Paraganglioma
Brief Title: Testing the Addition of an Anticancer Drug, Olaparib, to the Usual Chemotherapy (Temozolomide) for Advanced Neuroendocrine Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-03379; NCI-2020-03379 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); A021804 (Other: Alliance for Clinical Trials in Oncology); A021804 (Other: CTEP); U10CA180821 (NIH)
Record Dates: First submitted 2020-05-19; First posted 2020-05-20 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Advanced Adrenal Gland Pheochromocytoma; Advanced Paraganglioma; Metastatic Adrenal Gland Pheochromocytoma; Metastatic Paraganglioma; Stage III Adrenal Gland Pheochromocytoma and Sympathetic Paraganglioma AJCC v8; Stage IV Adrenal Gland Pheochromocytoma and Sympathetic Paraganglioma AJCC v8; Unresectable Adrenal Gland Pheochromocytoma; Unresectable Paraganglioma
MeSH Terms: conditions — Pheochromocytoma; Paraganglioma | interventions — Specimen Handling; Contrast Media; Magnetic Resonance Spectroscopy; olaparib; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (temozolomide, olaparib) (Experimental): Patients receive temozolomide PO QD and olaparib PO BID on days 1-7. Treatment with temozolomide repeats every 21 days for up to 13 cycles in the absence of disease progression or unacceptable toxicity. Cycles of olaparib repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo CT with contrast or MRI throughout the study and undergo mandatory collection of blood samples prior to treatment. Patients may optionally undergo collection of blood samples at the time of progression.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography with Contrast; Procedure: Magnetic Resonance Imaging; Drug: Olaparib; Other: Quality-of-Life Assessment; Drug: Temozolomide
- Arm II (temozolomide) (Active Comparator): Patients receive temozolomide PO QD on days 1-5. Treatment repeats every 28 days for up to 13 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo CT with contrast or MRI throughout the study and undergo mandatory collection of blood samples prior to treatment. Patients may optionally undergo collection of blood samples at the time of progression.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography with Contrast; Procedure: Magnetic Resonance Imaging; Other: Quality-of-Life Assessment; Drug: Temozolomide

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography with Contrast — Undergo CT with contrast
  Other Names: Contrast Enhanced Computed Tomography; CONTRAST ENHANCED CT SCAN; Contrast-enhanced Computed Tomography; CT Scan With Contrast; CT with Contrast
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Olaparib — Given PO
  Other Names: AZD 2281; AZD-2281; AZD2281; KU 0059436; KU-0059436; KU0059436; Lynparza; Olanib; Olaparix; PARP Inhibitor AZD2281
  Arms: Arm I (temozolomide, olaparib)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Gliotem; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temizole; Temodal; Temodar; Temomedac; TMZ

SUMMARY:
This phase II trial studies how well the addition of olaparib to the usual treatment, temozolomide, works in treating patients with neuroendocrine cancer (pheochromocytoma or paraganglioma) that has spread from where it first started (primary site) to other places in the body (metastatic) or cannot be removed by surgery (unresectable). Poly (adenosine diphosphate [ADP]-ribose) polymerases (PARPs) are proteins that help repair deoxyribonucleic acid (DNA) mutations. PARP inhibitors, such as olaparib, can keep PARP from working, so tumor cells can't repair themselves, and they may stop growing. Chemotherapy drugs, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving olaparib with temozolomide may shrink or stabilize the cancer in patients with pheochromocytoma or paraganglioma better than temozolomide alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the progression-free survival (PFS) of patients with advanced pheochromocytoma and paraganglioma (APP) receiving temozolomide (dose dense) and olaparib to that of patients receiving temozolomide (pulse dose) alone.

SECONDARY OBJECTIVES:

I. To compare the overall survival (OS) of patients with APP receiving temozolomide (dose dense) and olaparib versus (vs.) temozolomide (pulse dose) alone.

II. To compare the objective response rate (ORR) associated with temozolomide (dose dense) and olaparib vs. temozolomide (pulse dose) alone in patients with APP.

III. To evaluate and compare the toxicity profile of temozolomide-based combinations (temozolomide [dose dense] and olaparib vs. temozolomide [pulse dose]) in patients with APP using Common Terminology Criteria for Adverse Events (CTCAE) and Patient-Reported Outcomes (PRO)-CTCAE.

OTHER OBJECTIVE:

I. Results of the primary analysis will be examined for consistency, while taking into account the stratification factors and/or covariates of baseline quality of life (QOL) and fatigue.

EXPLORATORY OBJECTIVES:

I. To assess biochemical response: serum catecholamines and metanephrines; urine catecholamines and metanephrines.

II. To assess biomolecular markers associated with clinical outcome: germline succinyl dehydrogenase (SDH) mutations and tumor status of the repair enzyme methylguanine-deoxyribonucleic acid (DNA) methyltransferase (MGMT).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive temozolomide orally (PO) once daily (QD) and olaparib PO twice daily (BID) on days 1-7. Treatment with temozolomide repeats every 21 days for up to 13 cycles in the absence of disease progression or unacceptable toxicity. Cycles of olaparib repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo computed tomography (CT) with contrast or magnetic resonance imaging (MRI) throughout the study and undergo mandatory collection of blood samples prior to treatment. Patients may optionally undergo collection of blood samples at the time of progression.

ARM II: Patients receive temozolomide PO QD on days 1-5. Treatment repeats every 28 days for up to 13 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo CT with contrast or MRI throughout the study and undergo mandatory collection of blood samples prior to treatment. Patients may optionally undergo collection of blood samples at the time of progression.

Patients discontinuing treatment due to reasons other than disease progression are followed every 8 weeks until disease progression, then every 6 months until 5 years after start of treatment. Patients discontinuing treatment due to disease progression are followed every 6 months for 5 years after start of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of disease

  * Histologic documentation: Histologically-proven advanced (metastatic or unresectable primary) pheochromocytoma or paraganglioma
  * Stage: Advanced (metastatic or unresectable primary) disease
  * Tumor site: Histologically-proven pheochromocytoma or paraganglioma
  * Radiographic evaluation: Radiographic evidence of disease progression by Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1 in the 12 months prior to registration
* Measurable disease

  * Lesions must be accurately measured in at least one dimension (longest diameter to be recorded) as >= 1 cm with CT or MRI (or >= 1.5 cm for lymph nodes). Non-measurable disease includes disease smaller than these dimensions or lesions considered truly non-measurable including: leptomeningeal disease, ascites, pleural or pericardial effusion, lymphangitic involvement of skin or lung
* Prior treatment with other somatostatin analog, chemotherapy, radiotherapy (including peptide radionuclide receptor therapy [PRRT]), or surgery must be completed >= 28 days prior to registration. Patients must have recovered from any effects of any major surgery prior to registration
* Prior treatment with radiolabeled metaiodobenzylguanidine (MIBG) must be completed >= 12 weeks prior to registration and lifetime cumulative 131I-MIBG dose must be < 1000 MBq kg^-1 (36 mCi kg^-1)
* Prior treatment with antibiotics must be completed >= 7 days prior to registration
* No prior treatment with temozolomide, dacarbazine, or a poly ADP ribose polymerase (PARP) inhibitor
* No prior allogeneic bone marrow transplant or double umbilical cord blood transplantation (dUCBT)
* Not pregnant and not nursing, because this study involves an agent that has known genotoxic, mutagenic, and teratogenic effects. Therefore, for women of childbearing potential only, a negative pregnancy test done =< 7 days prior to registration is required
* Contraception

  * Therapy utilized in this trial is associated with medium/high fetal risk
  * Women of childbearing potential and their partners, who are sexually active, must agree to use two highly effective forms of contraception in combination. This should be started from the time of registration and continue throughout the period of taking study treatment and for at least 1 month after last dose of study drug(s), or they must totally/truly abstain from any form of sexual intercourse
  * Male patients must use a condom during treatment and for 3 months after the last dose of study drug(s) when having sexual intercourse with a pregnant woman or with a woman of childbearing potential. Female partners of male patients should also use a highly effective form of contraception if they are of childbearing potential. Male patients should not donate sperm throughout the period of taking study drug(s) and for 3 months following the last dose of study drug(s)
* Age >= 12 years
* Eastern Cooperative Oncology Group (ECOG) Patients ≥ 18 years of age: Performance status: 0-2

  * Patients < 16 years of age: Lansky ≥ 50%
  * Patients 16 to < 18 years of age: Karnofsky ≥ 50%
  * Patients ≥ 18 years of age: ECOG performance status ≤ 2
* Absolute neutrophil count >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Hemoglobin >= 10 mg/dL if prior radionuclide therapy Hemoglobin >= 8 mg/dL if no prior radionuclide therapy

  * In the absence of transfusion within the previous 24 hours. Radionuclide therapy includes PRRT or MIBG
* Total bilirubin =< 1.5 x upper limit of normal (ULN)

  * Except in the case of Gilbert's syndrome, then total bilirubin must be =< 3.0 x ULN
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 3.0 x ULN
* Creatinine < 1.5 x ULN OR calculated (calc.) creatinine clearance > 50 mL/min

  * Calculated by Cockcroft-Gault equation
  * By Cockcroft-Gault equation. Alternatively, for patients < 18 years of age, maximum serum creatinine ≤ the below age-sex-specific norms:

    * Age 12 years: Male 1.2; female 1.2
    * Age 13 to < 16 years: Male 1.5; female 1.4
    * Age 16 to < 18 years: Male 1.7; female 1.4
* No indication of uncontrolled, potentially reversible cardiac condition(s) as determined by investigator (e.g., unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, Fridericia's formula-corrected QT interval [QTcF] prolongation > 500 msec, electrolyte disturbances, etc.) and no known congenital long QT syndrome
* No extensive bilateral lung disease or pneumonitis
* No abnormal organ or bone marrow function =< 28 days prior to registration
* Patients with human immunodeficiency virus (HIV) positivity are allowed if CD4 count > 250 cells/uL and they have an undetectable HIV viral load within 6 months of registration
* No active infection
* No history of myelodysplastic syndrome (MDS) (or any dysplastic leukocyte morphology suggestive of MDS) or acute myeloid leukemia
* No known gastrointestinal condition(s) that might predispose for drug intolerability or poor drug absorption
* No known medical condition causing an inability to swallow oral formulations of agents
* No history of allergic reaction attributed to compounds of similar chemical or biologic composition to PARP inhibitors
* Concurrent use of combination antiretroviral therapy (ART) is not permitted
* Chronic concomitant treatment with strong or moderate CYP3A4 inducers or inhibitors is not allowed. Patients must discontinue the agent(s) >= 21 days prior to registration; enzalutamide and/or phenobarbital must be discontinued >= 5 weeks prior to registration

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-03-17 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From randomization to the first documentation of disease progression (per Response Evaluation Criteria in Solid Tumors [RECIST] version 1.1) or death, assessed up to 5 years
  Will be compared between treatment arms using the un-stratified log-rank test at one-sided level of 0.11 and the p-value will be used for decision making. The hazard ratio will be estimated using a Cox proportional hazards model and the 95% confidence interval for the hazard ratio will be provided. Results from a stratified analysis will also be provided. Kaplan-Meier methodology will be used to estimate the median PFS for each treatment arm, and Kaplan-Meier curves will be produced. Brookmeyer-Crowley methodology will be used to construct the 95% confidence interval for the median PFS for each treatment arm.

SECONDARY OUTCOMES:
Overall survival (OS) | From randomization to death due to any cause, assessed up to 5 years
  Patients who are alive will be censored at last follow-up. The distribution of survival time will be estimated using the method of Kaplan-Meier. OS will be compared between treatment arms using the log-rank test. OS medians, survival rates and hazard ratio will be estimated along with 95% confidence intervals.
Objective response | Up to 5 years
  Will be assessed by RECIST version 1.1 criteria. Will be estimated using objective response rate where objective response rate is defined as the number of evaluable patients achieving a response (partial response or complete response per RECIST version 1.1) during treatment with study therapy divided by the total number of evaluable patients. Rates of response will be compared across arms using a Chi-Square Test for Proportion. Point estimates will be generated for objective response rates within each arm along with 95% binomial confidence intervals.
Incidence of adverse events | Up to 5 years
  Will be assessed per National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The term toxicity is defined as adverse events that are classified as possibly, probably, or definitely related to study treatment. Toxicities will be evaluated via the ordinal Common Terminology Criteria for Adverse Events standard toxicity grading. Similarly, scores (0-4) and the maximum score for each Patient-Reported Outcomes-CTCAE item will be recorded for each patient.

OTHER OUTCOMES:
Biochemical response | Up to 5 years
  Levels of chromogranin A, urine and/or plasma catecholamines and metanephrines may predict response to therapy. The proportion of patients with a biochemical response of partial response or better, as determined by plasma and/or urine catecholamines and metanephrines, will be calculated, and a 95% confidence interval will be placed on this proportion. For each factor, we will calculate the mean +/- standard deviation, minimum, maximum, and quartiles; in addition, we will generate box and whisker plot.
Biomolecular markers associated with clinical outcome | Up to 5 years
  Will analyze for methyltransferase (MGMT) methylation expression in archival tumors and correlate with the radiographic response rate in metastatic pheochromocytoma/paraganglioma. This is hypothesis generated box and whisker plot.

CONTACTS AND LOCATIONS:
Overall Officials: Jaydira Del Rivero, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (163):
- United States (163):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber Cancer Institute - Chestnut Hill, Newton, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Henry Ford Saint John Hospital - Academic, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Breast, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Henry Ford Warren Hospital - Breast Macomb, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Henry Ford Rochester Hospital, Rochester Hills, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Madison Heights Hospital - Breast, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Albany Medical Center, Albany, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Farmington Health Center, Farmington, Utah
  - University of Utah Sugarhouse Health Center, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm